CLINICAL TRIAL: NCT04466917
Title: A Randomized, Double-blind, Phase 3 Bridging Study Evaluating the Safety and Efficacy of ABP 215 Compared With Bevacizumab in Chinese Subjects With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of ABP 215 Versus Bevacizumab in Chinese Subjects With Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to early terminate the study
Sponsor: Amgen (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20180085
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Non-small Cell Lung Cancer (NSCLC); Non-squamous NSCLC
Keywords: Biosimilar; Bevacizumab; Carboplatin; Paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive ABP 215 or bevacizumab on a 1:1 basis. All subjects will receive chemotherapy, following administration of investigational product.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, Amgen, designated PAREXEL, and other clinical site staff will be blinded to the investigational product allocation for each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABP 215 (Experimental): Subjects will be randomized to receive ABP 215 every 3 weeks (Q3W) for 6 cycles.
  All subjects will receive carboplatin and paclitaxel after the ABP 215 IV infusion every Q3W for at least 4 and not more than for 6 cycles.
  Interventions: Drug: ABP 215; Drug: Paclitaxel; Drug: Carboplatin
- Bevacizumab (Active Comparator): Subjects will be randomized to receive Bevacizumab every 3 weeks (Q3W) for 6 cycles.
  All subjects will receive carboplatin and paclitaxel after the Bevacizumab IV infusion every Q3W for at least 4 and not more than for 6 cycles.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: ABP 215 — ABP 215 will be administered at a dose of 15 mg/kg IV
  Arms: ABP 215
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg IV
  Arms: Bevacizumab
Drug: Paclitaxel — Paclitaxel will be administered 175 mg/m2 IV
Drug: Carboplatin — Carboplatin will be administered at an area under the concentration-time curve (AUC) of 5 IV

SUMMARY:
The purpose of this research study is to assess the efficacy and safety of ABP 215 compared to Bevacizumab in Chinese patients with advanced non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Approximately 170 subjects will be randomized 1:1 in approximately 40 sites in China. This study consists of a screening period of up to 28 days, followed by a treatment period of 18 weeks, and an end of study visit 3 weeks after the last dose of investigational product or study-specified chemotherapy. After randomization, subjects will receive investigational product at a dose of 15 mg/kg administered every 3 weeks for 6 cycles followed by at least 4 and no more than 6 cycles of carboplatin and paclitaxel chemotherapy every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-squamous NSCLC.
* Subjects must be initiating first-line carboplatin/paclitaxel chemotherapy within 8 days after randomization and expected to receive at least 4 and no more than 6 cycles of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Small cell lung cancer (SCLC) or mixed SCLC and NSCLC.
* Central nervous system (CNS) metastases.
* Malignancy other than NSCLC.
* Palliative radiotherapy for bone lesions inside the thorax.
* Prior radiotherapy of bone marrow.
* Active hepatitis B.
* Active hepatitis C.
* Tested positive for human immunodeficiency virus (HIV).
* Life expectancy < 6 months.
* Woman of childbearing potential who is pregnant or is breast feeding.
* Woman of childbearing potential who is not consenting to use highly effective methods of birth control during treatment and for an additional 6 months after the last administration of the protocol specified treatment.
* Man with a partner of childbearing potential who does not consent to use highly effective methods of birth control during treatment and for an additional 6 months after the last administration of the protocol specified treatment.
* Other exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-11-13 (Estimated); Study Completion 2022-11-13 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From Day 1 to Week 19 (EOS)
  The percentage of subjects with a best overall tumor response of Complete Response (CR) or Partial Response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From Day 1 to Week 19 (EOS)
Duration of response (DOR) | From Day 1 to Week 19 (EOS)
Maximum Plasma Concentration (Cmax) | Pre-dose on Week 1, Week 4, Week 7, Week 13 and Week 19 (EOS)
Area Under the Curve (AUC) | Pre-dose on Week 1, Week 4, Week 7, Week 13 and Week 19 (EOS)
Minimum observed concentration (Cmin) | Pre-dose on Week 1, Week 4, Week 7, Week 13 and Week 19 (EOS)
Number of participants with treatment-emergent adverse events | From Screening to Week 19 (EOS)
Number of participants with treatment-emergent events of interest (EOIs) | From Screening to Week 19 (EOS)
Number of participants with incidence of anti-drug antibodies (ADAs) | On Week 1, Week 7, Week 13 and Week 19 (EOS)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com